CLINICAL TRIAL: NCT01389648
Title: The Effect of Pre-operative Chest Physiotherapy on Post-operative Complications After Major Abdominal Surgery.
Brief Title: Pre-operative Physiotherapy to Prevent Post-operative Complications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: physiotherapyCTIL
Record Dates: First submitted 2011-07-06; First posted 2011-07-08 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2013-09

CONDITIONS: Abdominal Surgery
Keywords: adult
MeSH Terms: interventions — Preoperative Exercise

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pre Operative (Experimental): Pre operative chest physiotherapy treatment
  Interventions: Other: Pre Operative
- usual care (No Intervention)

INTERVENTIONS:
Other: Pre Operative — Pre operative chest physiotherapy treatment
  Arms: Pre Operative

SUMMARY:
The purpose of this study is to assess the roll of pre-operative chest physiotherapy, in addition to the usual care given after major abdominal surgery, in the prevention of post-operative respiratory complications.

ELIGIBILITY:
Inclusion Criteria:

* Major abdominal surgery

Exclusion Criteria:

* Respiratory Disease
* Pregnancy
* Mental Disease
* Dementia
* Alzheimer's Disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2011-11; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
respiratory complications | 6 months
  pneumonia, atelectasis

CONTACTS AND LOCATIONS:
Overall Officials: Yoram Kluger, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Health Care Campus, Haifa, Israel